CLINICAL TRIAL: NCT06547463
Title: Effects of Nasal Airflow on Sleep in Tracheotomized Patients
Acronym: Nasa
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240636
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Patients With Prolonged Weaning
Keywords: tracheostomy; sleep; nasal airflow

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with prolonged weaning: Mechanically ventilated tracheotomized patients admitted for ventilation weaning.
  Interventions: Other: nasal oxygenation device

INTERVENTIONS:
Other: nasal oxygenation device — Use of the nasal oxygenation device on one of the two nights during which polysomnography will be performed.

SUMMARY:
The passage of air through the nasal cavities generates rhythmic oscillations transmitted by the olfactory bulb to the brain, which induces cerebral activation in functional brain areas and is associated with better cognitive performance compared to oral breathing. Consequently, the abolition of nasal ventilation - intrinsic in tracheotomized and ventilated patients - could have deleterious effects on brain activity. Besides the loss of olfaction, the abolition of nasal ventilation could affect brain activity and sleep.

The hypothesis of the present study is that the restoration of nasal stimulation by the passage of humidified nasal airflow in tracheotomized and ventilated patients improves sleep quality, notably with a greater proportion of time spent in REM sleep.

DETAILED DESCRIPTION:
The use of invasive mechanical ventilation via an endotracheal tube or tracheotomy involves bypassing the nasopharyngeal space and abolishing nasal ventilation. The first consequence is the loss of olfactory function. This function is quickly recovered when nasal ventilation is made possible. However, the abolition of nasal ventilation may have consequences beyond the loss of olfaction. The abolition of nasal ventilation in intubated rats inhibits these rhythmic oscillations, which can be restored by nasal sprays. In humans, nasal ventilation induces cerebral activity in functional brain areas and is associated with better cognitive performance compared to oral ventilation. In a model of intubated and ventilated rats, it has been shown that nasal sprays synchronized with the ventilator reduce hippocampal lesions compared to animals ventilated with an endotracheal tube without nasal sprays. Finally, in patients intubated with an endotracheal tube for toxic comas, the same nasal spray system restored brain activity and neural connectivity.

The aim of this study is to test the effects of nasal airflow of the sleep in tracheostomized patients who are still dependent to invasive mechanical ventilation. Patients will be investigated by a full polysomnography during two consecutive nights, with and without nasal airflow on the top of invasive mechanical ventilation, the two nights being randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Admission to PRRS for weaning from ventilation
3. Tracheotomy and nocturnal invasive mechanical ventilation
4. Indication for polysomnography by care team
5. Agreement to participate by patient or trusted person/relative and signature of consent form
6. Affiliation with a social security scheme or beneficiary

Exclusion Criteria:

1. Diseases of the central nervous system: cerebrovascular accident (CVA), multiple sclerosis (MS), epilepsy
2. Psychiatric illnesses (psychoses)
3. Hyperthermia (temperature > 38.5°C)
4. Agitation, resuscitation delirium
5. Continuous use of sedatives
6. Patients under legal protection (guardianship/curatorship)
7. Patients deprived of liberty by judicial or administrative decision
8. Patients under AME
9. Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated tracheotomized patients admitted for ventilation weaning.
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-04-13 (Estimated); Study Completion 2026-04-13 (Estimated)

PRIMARY OUTCOMES:
Effects of nasal ventilation on sleep quality in ventilation-dependent tracheostomized patients. | During the 12 hours duration of PSG
  The proportion of time spent in REM sleep over the total sleep time

SECONDARY OUTCOMES:
Effects of nasal ventilation on sleep duration | During the 12 hours duration of PSG
  Total sleep time as determined by polysomnography
Effects of nasal ventilation on sleep architecture | During the 12 hours duration of PSG
  Proportion of time spent in stage 1, stage 2 and stage 3 sleeping
Effects of nasal ventilation on the proportion of atypical sleep | During the 12 hours duration of PSG
  Proportion of time spent in atypical sleep
Effects of nasal ventilation on minute ventilation | During the 12 hours duration of PSG
  Measurement of transcutaneous PaCO2
Effects of nasal ventilation on night-time awakenings | During the 12 hours duration of PSG
  Prevalence of night-time awakenings
Effects of nasal ventilation on patient-ventilator asynchrony | During the 12 hours duration of PSG
  Asynchrony index (number of asynchronies/total number of respiratory cycles)

CONTACTS AND LOCATIONS:
Locations (1):
- Pitié Salpétrière HOSPITAL, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal